CLINICAL TRIAL: NCT07060092
Title: Network Analysis of Bodywide Coordination Supporting Suprapostural Dexterity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0055-23-EP
Record Dates: First submitted 2025-06-25; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Trail Making Task; Balance Board
Keywords: Movement disorder; Postural instability; Fall prevention; Dexterity; Suprapostural control; Motor coordination; Whole-body coordination; Multiplicative interactions; Modular motor networks; Nonlinear movement variability; Trail Making Test (TMT); Posturography; Whole-body kinematics; Eye tracking; Network analysis; Rehabilitation science
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Intervention Model Description: This is a within-subject, factorial study investigating how suprapostural dexterity emerges from multiplicative interactions across the human movement system under varying task demands and surface stability conditions. Fifty healthy adults will complete a series of upright standing and whole-body Trail Making Test tasks on stable and unstable surfaces while posturography, full-body kinematics, and eye tracking data are recorded and analyzed using multifractal and network modeling techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trail Making Task on Stable Surface (Experimental): Participants perform the Trail Making Task while standing on stable force plates.
  Interventions: Behavioral: Trail Making Task
- Standing on Unstable Surface (Experimental): Participants maintain upright stance on a balance board placed atop force plates (no cognitive task).
  Interventions: Behavioral: Balance board
- Trail Making Task on Unstable Surface (Experimental): Participants perform the Trail Making Task while standing on a balance board, requiring simultaneous postural and cognitive-motor coordination.
  Interventions: Behavioral: Trail Making Task; Behavioral: Balance board

INTERVENTIONS:
Behavioral: Trail Making Task — Participants will perform a modified, life-size version of the Trail Making Test (TMT) while standing upright, either on a stable (force plates) or unstable (balance board) surface. The task involves visually searching for and tracing a sequential path through spatially randomized numerical targets projected onto a large screen using a laser pointer. This dual-task condition simultaneously engages cognitive, visual, and motor planning systems while requiring continuous postural control. The task is designed to elicit suprapostural coordination, capturing the dynamic interplay between postural stability and goal-directed behavior.
  Arms: Trail Making Task on Stable Surface; Trail Making Task on Unstable Surface
Behavioral: Balance board — Participants will maintain an upright stance on a commercially available balance board positioned atop dual force plates. The unstable surface introduces controlled postural instability, requiring continuous sensorimotor adaptation to preserve balance without external support. This condition is administered alone and in combination with the Trail Making Task to simulate dual-task challenges that more closely resemble real-world balance demands.
  Arms: Standing on Unstable Surface; Trail Making Task on Unstable Surface

SUMMARY:
Prevailing understandings of movement disorders characterize "broken" movements in a piecewise fashion, for instance, focusing on motor control, muscle tone, posture, or cognition independently of each other. These fractured approaches to movement coordination are blind to the body's functional integrity. Consequently, rehabilitative interventions target the limb or body parts most affected by the disorder, seeking to support the whole body by mending the broken part. However, dexterity is global, functional coordination spanning the whole body. In other words, task completion draws on fundamental interactivity, allowing the body to coordinate various anatomical parts. This coordination may be more vital to healthy movement than individual anatomical parts. Understanding this interactivity is thus paramount to developing novel rehabilitative interventions to prevent falls and improve the quality of life in pathological populations. Studying bodywide coordination for suprapostural dexterity requires innovation in experimental setup and analytical techniques. This project integrates a customizable life-size Trail Making Test with posturography, whole-body movement tracking, eye tracking, and state-of-the-art cascade modeling and network analysis methods to assess functional coordination across the whole body. The experimenters will leverage causal network analyses of multiplicative interactions instrumental in previous studies of whole-body exploratory motor behavior but not yet utilized in studying suprapostural dexterity. Aim 1 will investigate how multiplicative interactions among movement-system components support suprapostural dexterity. The experimenters hypothesize that maintaining an upright stance would produce a functional network of multiplicative interactions among movement-system components. The experimenters also hypothesize that participating in the Trail Making Test would produce a succession of distinct, modular networks of multiplicative interactions among movement-system components. Aims 2 will investigate how multiplicative interactions among movement-system components support suprapostural dexterity in the face of postural instability. The experimenters hypothesize that destabilizing contact with the ground surface when maintaining an upright stance will produce modular networks of multiplicative interactions with increased connectivity among these modules compared to stable standing. The experimenters also hypothesize that destabilizing contact with the ground surface in the Trail Making Test would produce a succession of distinct, modular networks of multiplicative interactions with increased connectivity among these modules compared to stable standing. This modeling framework offers a new way to understand suprapostural dexterity and its breakdown in various movement disorders in light of recent theoretical developments in cascade modeling and network physiology.

DETAILED DESCRIPTION:
It is estimated that 42 million people in the United States might suffer from some form of movement disorder. Prevailing understandings of these movement disorders characterize "broken" movements in a piecewise fashion, for instance, focusing on motor control, muscle tone, posture, or cognition independently of each other. These fractured approaches to movement coordination are blind to the body's functional integrity. Consequently, rehabilitative interventions target the limb or body parts most affected by the disorder seeking to support the whole body by mending the broken part. However, dexterity is global, functional coordination spanning the whole body. Suprapostural dexterity, for instance, when the task requires an upright posture, is a prime example of how functionality can triumph over anatomical separability. Whatever starts at one or more anatomical areas can swiftly spread throughout the entire body, destabilizing the body on the potential path to task completion. In individuals with movement disorders, the impaired coordination between task engagement and postural instability amplifies the risk of falling. Developing novel rehabilitative interventions to prevent falls and improve the quality of life in individuals with movement disorders thus requires understanding how task completion depends on essential interaction that enables the body to coordinate different anatomical parts.

This project investigates how multiplicative interactions support suprapostural dexterity from two complementary premises. First, movement science has established that postural stability requires a modular structure of functional networks shaped by anatomical constraints. This arrangement indicates a soft assembly and disassembly of functional modules as an individual engages in a task and responds to changing task demands, respectively. Second, movement science has yet to grapple with the multiplicative interactions among movement-system components producing highly complex and unpredictable behaviors beyond the scope of dominant linear modeling approaches. The scientific premises for this proposal are that the dominant network approaches to dexterity are linear, and network approaches can give voice to the nonlinearity we all know is there.

Studying multiplicative interactions among movement-system components and suprapostural dexterity requires innovation in experimental setup and analytical techniques. This project integrates a customizable life-size Trail Making Test (TMT) with posturography, whole-body movement tracking, and eye tracking, along with state-of-the-art cascade modeling and network analysis methods to assess functional coordination across the whole body. The experimenters will leverage causal network analyses of multiplicative interactions instrumental in previous studies of whole-body exploratory motor behavior but not yet utilized in studying suprapostural dexterity.

Specific Aim 1: To investigate how multiplicative interactions among movement-system components support suprapostural dexterity.

Hypothesis 1.1: The experimenters hypothesize that maintaining an upright stance would produce a functional network of multiplicative interactions among movement-system components.

Hypothesis 1.2: The experimenters hypothesize that participating in the Trail Making Test would produce a succession of distinct, modular networks of multiplicative interactions among movement-system components.

Specific Aim 2: To investigate how multiplicative interactions among movement-system components support suprapostural dexterity in the face of postural instability.

Hypothesis 2.1: The experimenters hypothesize that destabilizing contact with the ground surface when maintaining an upright stance will produce modular networks of multiplicative interactions with increased connectivity among these modules compared to stable standing.

Hypothesis 2.2: The experimenters hypothesize that destabilizing contact with the ground surface in the Trail Making Test would produce a succession of distinct, modular networks of multiplicative interactions with increased connectivity among these modules compared to stable standing.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide informed consent
* Be able to stand and walk independently without an assistive device

Exclusion Criteria:

* Self-report any diagnosis of a neurological disease
* Self-report any diagnosis of any limb disabilities, injuries, or disease.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Network structure | Day 1
  The outcome measure characterizes the directional, weighted network of multiplicative interactions across the human movement system, derived from vector autoregression (VAR) analysis of multifractal fluctuations in center-of-pressure (CoP), center-of-mass (CoM), and 79 anatomical marker displacement series. Each node in the network represents a body segment or anatomical location, and each edge captures the strength and direction of influence in nonlinear fluctuation propagation across time. These networks are modeled individually for each participant and task condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Biomechanics Research Building, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT07060092/Prot_000.pdf